CLINICAL TRIAL: NCT05014087
Title: Digoxin In Treatment of Alcohol Associated Hepatitis (DIGIT-AlcHep)
Brief Title: Digoxin In Treatment of Alcohol Associated Hepatitis
Acronym: DIGIT-AlcHep
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Bubu Banini, MD, PhD, Assistant Professor of Internal Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000030659
Record Dates: First submitted 2021-07-20; First posted 2021-08-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Acute Alcoholic Hepatitis; Chemical and Drug Induced Liver Injury; Alcohol-Induced Disorders; Steatohepatitis Caused by Ingestible Alcohol
Keywords: Acute alcoholic hepatitis; Liver injury; Liver inflammation; Liver disease; Digoxin
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Alcohol-Induced Disorders; Fatty Liver, Alcoholic; Hepatitis; Liver Diseases | interventions — Digoxin

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open label, randomized 1:1 controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Digoxin (Experimental): In the digoxin arm, the intervention to be administered will be intravenous digoxin dosed by weight and by renal function using an adaption of the established FDA nomogram. Participants randomized to digoxin will receive an intravenous digoxin loading dose administered in 3 doses over 24 hours starting on Day 1. Digoxin levels will be monitored daily throughout the participant's hospital stay, to a maximum of 28 days. Digoxin will be discontinued at the time discharge if before 28 days.
  Interventions: Drug: Intravenous digoxin
- Arm B: No Digoxin (No Intervention): In the no digoxin arm, no study drug or placebo will be administered.

INTERVENTIONS:
Drug: Intravenous digoxin — Loading dose: the total loading dose of digoxin will be determined using the Loading nomogram. The FDA-recommended total IV digoxin loading dose range is 8 to 12 mcg/kg. The lowest recommended dose of 8 mcg/kg was used in constructing the digoxin Loading nomogram that will be used in this trial.
  Maintenance dose: the maintenance dose will be started approximately 24 hours after initiation of digoxin loading. The post-loading digoxin trough will be reviewed prior to starting maintenance dosing.
  Subjects on P-gp inhibitors or spironolactone, will have an additional digoxin level performed 12-hours after any dose adjustment. Once digoxin levels are stable, 24-hour blood draws will be performed.
  Other Names: Lanoxin
  Arms: Arm A: Digoxin

SUMMARY:
Prospective, single center, open label, randomized controlled trial to explore whether digoxin treatment affects cytokine levels as biomarkers of inflammation in patients with acute alcohol associated hepatitis, digoxin administration and dose adjustment.

The study intervention will be intravenous digoxin (renal-based dosing for maximum of 28 days) versus no digoxin in an open-label 1:1 randomized allocation of patients with severe acute alcohol associated hepatitis.

DETAILED DESCRIPTION:
Severe alcohol associated hepatitis is a condition of acute on chronic immune liver dysfunction that is associated with high mortality, necessitating a search for drugs that may prove safe and efficacious in treating this disease. Pre-clinical studies suggest that digoxin, which is currently used for treating cardiac conditions, is also effective in improving alcohol-associated liver injury. To date, there have been no clinical studies of digoxin use in patients with alcohol associated hepatitis.

The primary objective of this randomized control study of digoxin versus no digoxin in patients with severe alcohol associated hepatitis is to explore whether digoxin treatment affects cytokine levels as biomarkers of inflammation in patients hospitalized with severe alcohol associated hepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of alcohol associated hepatitis based on clinical criteria or histologic evidence

1. Clinical criteria:

   * Onset of jaundice (bilirubin >3 mg/dL) within the prior 8 weeks
   * Regular alcohol use > 6 months, with intake of > 40 g/day (>280 g/week) for women; and > 60 g/day (>420 g/week) for men
   * AST > 50 IU/l
   * AST: ALT > 1.5 and both values < 400 IU/l
2. Histological evidence of alcohol associated hepatitis*

   2. MDF >32 or MELD ≥ 20 to ≤ 35 on Day 0 of the trial

   3. Age between 21 and 70 years, inclusive

   * In patients with possible alcohol associated hepatitis with confounding factors such as possible ischemic hepatitis, possible DILI, uncertain history of alcohol use, or atypical/abnormal laboratory tests (e.g., AST < 50 IU/IU/L or > 400 IU/IU/L, AST/ALT ratio < 1.5), antinuclearantibody > 1:160 or SMA > 1:80, standard of care liver biopsy may be performed as per discretion of the primary attending physician to confirm alcohol associated hepatitis and exclude competing etiologies. The decision to perform liver biopsy will be made by the primary team and will occur regardless of the study. As per current SOC, a liver biopsy may be obtained to confirm suspected alcohol-associated hepatitis and to rule out other potential etiologies of liver disease.

   If a liver biopsy is performed for clinically indicated reasons, we will store liver tissue that is left over after the portion needed for the primary indication has been identified.

   Exclusion Criteria:
   1. - Currently pregnant or breastfeeding
   2. - Inability of patient, legally authorized representative or next-of-kin to provide informed consent
   3. - Allergy or intolerance to digoxin
   4. - Clinically active C. diff infection
   5. - Positive test for COVID-19 within 14 days prior to the screening visit
   6. - Acute hepatitis E, Cytomegalovirus, Epstein Barr Virus, Herpes Simplex Virus

   7- History of other liver diseases including hepatitis B (positive HBsAg or HBV DNA), hepatitis 8-C (positive HCV RNA), autoimmune hepatitis, Wilson disease, genetic hemochromatosis, alpha1-antitrypsin deficiency.

   8-Diagnosis of Drug Induced Liver Injury (DILI), or other etiologies seen on liver imaging.

   9 - History of HIV infection (positive HIV RNA or on treatment for HIV infection)

   10 - Current diagnosis of cancer

   11- Renal failure defined by GFR <30 mL/min

   12 - Refractory ascites, defined as having more than 4 paracenteses in the preceding 8 weeks despite diuretic therapy

   13 - Prior exposure to experimental therapies or other clinical trial in last 3 months

   14 - Current acute or chronic pancreatitis

   15 - Active gastrointestinal bleeding unless resolved for >48 hours

   16 - Experiencing withdrawal seizures or considered at high risk for alcohol withdrawal seizures or delirium tremens

   17 - Heart rate less than 60 bpm at screening visit or at baseline

   18 - Current diagnosis of atrial fibrillation

   19 - Cardiomyopathy

   20 - Heart failure

   21 - Severe aortic valve disease

   22 - Presence of Accessory arterio-ventricular pathway (eg Wolf-Parkinson-White syndrome)

   23 - Complete heart block or second degree arterio-ventricular block without pacemaker or implantable cardiac device

   24 - Any of the following within the previous 6 months: myocardial infarction, percutaneous intervention, pacemaker/implantable cardiac device implantation, cardiac surgery or stroke

   25 - Current use of the following medications:
   * Antiarrhythmic (amiodarone, dofetilide, sotalol, dronedarone)
   * Parathyroid hormone analog (teriparatide)
   * Thyroid supplement (thyroid, levothyroxine sodium)
   * Sympathomimetics or ionotropic drugs (epinephrine, norepinephrine, dopamine, dobutamine, milrinone)
   * Neuromuscular blocking agents (succinylcholine)
   * Calcium supplement
   * Ivabradine
   * Disulfiram

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of inflammation | day 3
  Change in biomarkers of inflammation cytokine levels (pg/mL) in participants with acute alcohol associated hepatitis treated with digoxin versus no digoxin at day 3 of the study .

SECONDARY OUTCOMES:
Practicality of daily digoxin measurements | Up to 28 days
  Time to 90% of patients have digoxin checked levels within the pre-specified time window
Feasibility of digoxin dosing in a timely manner. | Up to 28 days
  Time to 90% of patients receive every scheduled dose of the drug
Feasibility of digoxin dose adjustments in renal insufficiency. | Up to 28 days
  90% of necessary dose adjustments were made appropriately in response to digoxin levels
Mortality at 7, 14, 28, 90 days. All cause mortality of patients enrolled in the trial. | Up to 90 days
  The mortality rates at different time points in the digoxin group and in the control group
Development of ECG abnormalities | Up to 28 days
  The number and proportion of patients in the digoxin and control groups with ECG changes compared to baseline
Recruitment | up to 90 days
  Ability to recruit 4 patients per month IS THIS A YES/NO or can we present it as the mean number of participants recruited per month?

OTHER OUTCOMES:
Organ dysfunction (Liver - Lille Score) | Up to 28 days
  Changes in liver-related function will be determined through assessment of Lille score. The model is based on: Age, Albumin, Bilirubin (initial), Bilirubin (day 7), Creatinine, PT. Survival probability at 6 months is defined by a cutoff of 0.45: 6-month survival probability of patients with a Lille model above 0.45 is about 25% contrary to patients with a Lille model below this cutoff (85% survival).
Organ dysfunction (Liver) with Model for End-stage Liver Disease (MELD) | Up to 28 days
  Changes in liver-related function will be determined through assessment of Model for End-stage Liver Disease (MELD) score, a number that ranges from 6 (least sick) to 40 (most sick) based on blood tests. The lab tests used to determine the MELD score are creatinine, bilirubin, sodium and international normalized ratio (INR).
Organ dysfunction (Liver Enzyme: Bilirubin) | Up to 28 days
  Changes in liver-related function will be determined through assessment of the liver enzyme bilirubin
Organ dysfunction (Liver Enzyme: Alkaline Phosphatase [ALP]) | Up to 28 days
  Changes in liver-related function will be determined through assessment of liver enzymes (alkaline phosphatase [ALP])
Organ dysfunction (Liver Enzyme: Aspartate Aminotransferase [AST]) | Up to 28 days
  Changes in liver-related function will be determined through assessment of liver enzymes (aspartate aminotransferase [AST])
Organ dysfunction (Liver Enzyme: Alanine Aminotransferase [ALT]) | Up to 28 days
  Changes in liver-related function will be determined through assessment of liver enzymes (alanine aminotransferase [ALT])
Organ Dysfunction (Multi-Organ) with Sequential Organ Failure Assessment (SOFA) | Up to 28 days
  Dysfunction in other organs will be assessed using Sequential Organ Failure Assessment (SOFA) score which is calculated based on a person's liver function, kidney function, nervous system, coagulation, circulation, and respiratory status. The score ranges from 0 (least sick) to 24 (most sick).
Organ Dysfunction (Multi-Organ) with the Multi-Organ Dysfunction Score (MODS) | Up to 28 days
  Dysfunction in other organs will be assessed using Multi-organ dysfunction score (MODS), calculated based on a person's liver function, kidney function, nervous system, coagulation, circulation, and respiratory status. The score ranges from 0 (least sick) to 24 (most sick).
Development of new or recurrent renal failure. | Up to 28 days
  Creatinine rise ≥ 0.5 mg/dL or ≥ 20% from baseline or requiring renal replacement therapy.
Racial and ethnic diversity in subject recruitment and retention. | Up to 90 days
  Race and ethnicity of enrolled subjects and subjects who completed the study will be summarized using count and proportion to assess the study's objective of enrolling and retaining at least 10% Black and at least 10% Hispanic participants to study completion (90-days follow-up)follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Bubu Banini, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maddrey WC, Boitnott JK, Bedine MS, Weber FL Jr, Mezey E, White RI Jr. Corticosteroid therapy of alcoholic hepatitis. Gastroenterology. 1978 Aug;75(2):193-9. PMID 352788
- [Background] Sahlman P, Nissinen M, Pukkala E, Farkkila M. Incidence, survival and cause-specific mortality in alcoholic liver disease: a population-based cohort study. Scand J Gastroenterol. 2016 Aug;51(8):961-6. doi: 10.3109/00365521.2016.1157889. Epub 2016 May 16. PMID 27181618
- [Background] Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, Downs N, Gleeson D, MacGilchrist A, Grant A, Hood S, Masson S, McCune A, Mellor J, O'Grady J, Patch D, Ratcliffe I, Roderick P, Stanton L, Vergis N, Wright M, Ryder S, Forrest EH; STOPAH Trial. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med. 2015 Apr 23;372(17):1619-28. doi: 10.1056/NEJMoa1412278. PMID 25901427
- [Background] Scalese MJ, Salvatore DJ. Role of Digoxin in Atrial Fibrillation. J Pharm Pract. 2017 Aug;30(4):434-440. doi: 10.1177/0897190016642361. Epub 2016 Apr 10. PMID 27067743
- [Background] Ouyang X, Han SN, Zhang JY, Dioletis E, Nemeth BT, Pacher P, Feng D, Bataller R, Cabezas J, Starkel P, Caballeria J, Pongratz RL, Cai SY, Schnabl B, Hoque R, Chen Y, Yang WH, Garcia-Martinez I, Wang FS, Gao B, Torok NJ, Kibbey RG, Mehal WZ. Digoxin Suppresses Pyruvate Kinase M2-Promoted HIF-1alpha Transactivation in Steatohepatitis. Cell Metab. 2018 Feb 6;27(2):339-350.e3. doi: 10.1016/j.cmet.2018.01.007. PMID 29414684
- [Background] Arteel GE, Iimuro Y, Yin M, Raleigh JA, Thurman RG. Chronic enteral ethanol treatment causes hypoxia in rat liver tissue in vivo. Hepatology. 1997 Apr;25(4):920-6. doi: 10.1002/hep.510250422. PMID 9096598
- [Background] Lee YS, Kim JW, Osborne O, Oh DY, Sasik R, Schenk S, Chen A, Chung H, Murphy A, Watkins SM, Quehenberger O, Johnson RS, Olefsky JM. Increased adipocyte O2 consumption triggers HIF-1alpha, causing inflammation and insulin resistance in obesity. Cell. 2014 Jun 5;157(6):1339-1352. doi: 10.1016/j.cell.2014.05.012. PMID 24906151
- [Background] Nath B, Levin I, Csak T, Petrasek J, Mueller C, Kodys K, Catalano D, Mandrekar P, Szabo G. Hepatocyte-specific hypoxia-inducible factor-1alpha is a determinant of lipid accumulation and liver injury in alcohol-induced steatosis in mice. Hepatology. 2011 May;53(5):1526-37. doi: 10.1002/hep.24256. PMID 21520168
- [Background] Palmer BF, Clegg DJ. Ascent to altitude as a weight loss method: the good and bad of hypoxia inducible factor activation. Obesity (Silver Spring). 2014 Feb;22(2):311-7. doi: 10.1002/oby.20499. Epub 2013 Oct 15. PMID 23625659
- [Background] Semenza GL. Hypoxia-inducible factors in physiology and medicine. Cell. 2012 Feb 3;148(3):399-408. doi: 10.1016/j.cell.2012.01.021. PMID 22304911
- [Background] Hollman A. Drugs for atrial fibrillation. Digoxin comes from Digitalis lanata. BMJ. 1996 Apr 6;312(7035):912. doi: 10.1136/bmj.312.7035.912. No abstract available. PMID 8611904
- [Background] Digoxin FDA insert. . [cited 2021 3/15/2021]
- [Background] (CDC)., C.f.D.C.a.P. Alcohol and Public Health: Alcohol-Related Disease Impact (ARDI). Annual Average for United States 2011-2015 Alcohol-Attributable Deaths Due to Excessive Alcohol Use, All Ages. [cited 2021 3/20/2021]
- [Background] (NIH)., N.I.o.H. Alcohol Facts and Statistics. [cited 2021 3/20/2021]
- [Background] Rathore SS, Curtis JP, Wang Y, Bristow MR, Krumholz HM. Association of serum digoxin concentration and outcomes in patients with heart failure. JAMA. 2003 Feb 19;289(7):871-8. doi: 10.1001/jama.289.7.871. PMID 12588271
- [Background] Ouyang AJ, Lv YN, Zhong HL, Wen JH, Wei XH, Peng HW, Zhou J, Liu LL. Meta-analysis of digoxin use and risk of mortality in patients with atrial fibrillation. Am J Cardiol. 2015 Apr 1;115(7):901-6. doi: 10.1016/j.amjcard.2015.01.013. Epub 2015 Jan 14. PMID 25660972
- [Background] Dasgupta A. Endogenous and exogenous digoxin-like immunoreactive substances: impact on therapeutic drug monitoring of digoxin. Am J Clin Pathol. 2002 Jul;118(1):132-40. doi: 10.1309/3VNP-TWFQ-HT9A-1QH8. PMID 12109847
- [Background] Yang SS, Hughes RD, Williams R. Digoxin-like immunoreactive substances in severe acute liver disease due to viral hepatitis and paracetamol overdose. Hepatology. 1988 Jan-Feb;8(1):93-7. doi: 10.1002/hep.1840080119. PMID 2828215
- [Background] Rosenkranz B, Frolich JC. Falsely elevated digoxin concentrations in patients with liver disease. Ther Drug Monit. 1985;7(2):202-6. doi: 10.1097/00007691-198506000-00011. PMID 4024214
- [Background] Nikou GC, Vyssoulis GP, Venetikou MS, Karga HI, Karoutsos KA, Toutouzas PK. Digoxin-like substance(s) interfere(s) with serum estimations of the drug in cirrhotic patients. J Clin Gastroenterol. 1989 Aug;11(4):430-3. doi: 10.1097/00004836-198908000-00016. PMID 2547866
- [Background] Digoxin conversion calculator.
- [Background] O'Shea RS, Dasarathy S, McCullough AJ; Practice Guideline Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Alcoholic liver disease. Hepatology. 2010 Jan;51(1):307-28. doi: 10.1002/hep.23258. No abstract available. PMID 20034030
- [Background] Bode C, Bode JC. Effect of alcohol consumption on the gut. Best Pract Res Clin Gastroenterol. 2003 Aug;17(4):575-92. doi: 10.1016/s1521-6918(03)00034-9. PMID 12828956
- [Background] Trial of Anakinra (Plus Zinc) or Prednisone in Patients With Severe Alcohol associated Hepatitis (AlcHepNet). [cited 2021 03/29]
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing 2020